CLINICAL TRIAL: NCT00123539
Title: Estradiol for Neurocognitive Dysfunction After CABG
Brief Title: Estrogen Replacement to Reduce Risk of Neurologic Injury After Coronary Artery Bypass Graft Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB stopped the study based on conclusion of likely futility of treatment on the primary outcome.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Charles W. Hogue, MD, The Johns Hopkins Medical Institutions
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 237; R01HL064600 (NIH)
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2007-12

CONDITIONS: Coronary Disease; Cardiovascular Diseases; Heart Diseases; Neurologic Manifestations
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Heart Diseases; Neurologic Manifestations | interventions — Estrogen Replacement Therapy; Surgical Procedures, Operative

INTERVENTIONS:
Drug: Estrogen Replacement Therapy
Procedure: Surgery

SUMMARY:
The purpose of this study is to test whether perioperative estrogen replacement in postmenopausal women reduces the risk for neurologic injury after coronary artery bypass graft (CABG) surgery.

DETAILED DESCRIPTION:
BACKGROUND:

Women undergoing CABG surgery have a higher operative mortality rate, longer hospitalizations, and higher hospital costs compared with men. A large proportion of this excess morbidity and mortality of surgery for women is due to perioperative neurologic injury. Estrogen has been consistently shown to reduce the extent of neurologic injury in a variety of in vitro and animal experimental stroke models. These data together strongly suggest that the higher risk for perioperative neurologic complications for elderly women may relate to their estrogen deficient state.

DESIGN NARRATIVE:

This randomized, placebo controlled study will test the hypothesis that perioperative estrogen replacement in postmenopausal women reduces the risk for neurologic injury after CABG surgery. Three hundred thirty-four women undergoing CABG surgery will be prospectively randomized to receive either 17 beta-estradiol or placebo in a double-blind fashion beginning the day before surgery and continuing for 5 days after surgery. Patients will be assessed for neurocognitive dysfunction, which is the most common manifestation of neurologic injury from cardiac surgery. Neurocognitive testing will be performed 1 to 2 days before surgery, 4 to 6 weeks postoperatively, and 6 months after surgery. The primary endpoint will be neurocognitive function 4 to 6 weeks after surgery for women who received 17 beta- estradiol compared with placebo perioperatively. The trial will also evaluate the importance of postoperative cognitive decline on measures of cognitive function and quality of life 6 months after surgery, and whether perioperative 17 beta-estradiol treatment improves these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose scheduled procedure is CABG surgery OR
* Patients whose scheduled procedure is isolated aortic surgery OR
* Patients whose scheduled procedure is mitral valve surgery OR
* Patients whose scheduled procedure is CABG combined with aortic or mitral valve surgery

Exclusion Criteria:

* Patients having re-operations
* Patients having combined carotid endarterectomy with CABG surgery
* Patients having CABG with tricuspid valve surgery
* Patients having mitral and aortic valvular surgery (with or without CABG surgery)
* Elevation of liver function test before surgery or creatinine before surgery greater than 2 mg/dl
* Emergency surgery
* Severe cognitive impairment before surgery as indicated by clinical history and/or a score greater than 12 on the Short Blessed Dementia Screening Test (see d11)
* Inability to attend outpatient visits
* A history of venous thromboembolism
* Unexplained vaginal bleeding
* A history of breast cancer or personal history of endometrial cancer in the absence of hysterectomy
* Estrogen use within 6 months of the surgery
* Patient refusal to participate
* Inability to speak and read English or visual impairment

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334
Dates: Start 2001-06; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Neurocognitive function (measured 4 to 6 weeks after surgery)
Cognitive function
Quality of life (measured 6 months after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Charles W. Hogue, Jr., MD, Principal Investigator — Department of Anesthesiology and Critical Care Medicine, The Johns Hopkins University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Stearns JD, Davila-Roman VG, Barzilai B, Thompson RE, Grogan KL, Thomas B, Hogue CW Jr. Prognostic value of troponin I levels for predicting adverse cardiovascular outcomes in postmenopausal women undergoing cardiac surgery. Anesth Analg. 2009 Mar;108(3):719-26. doi: 10.1213/ane.0b013e318193fe73. PMID 19224775
- [Derived] Hogue CW, Fucetola R, Hershey T, Freedland K, Davila-Roman VG, Goate AM, Thompson RE. Risk factors for neurocognitive dysfunction after cardiac surgery in postmenopausal women. Ann Thorac Surg. 2008 Aug;86(2):511-6. doi: 10.1016/j.athoracsur.2008.04.058. PMID 18640325